CLINICAL TRIAL: NCT00576251
Title: TOBRADEX Ophthalmic Suspension Versus Tobramycin 0.3%/Dexamethasone 0.05% Ophthalmic Suspension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Judy Vittitoe, Alcon Research
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-07-19
Record Dates: First submitted 2007-12-17; First posted 2007-12-19 (Estimated); Results first posted 2010-01-14 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-02

CONDITIONS: Ocular Inflammation Associated With Blepharaconjunctivitis
Keywords: Ocular inflammation; blepharaconjunctivitis
MeSH Terms: interventions — Tobramycin; Tobramycin, Dexamethasone Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tobramycin 0.3%/Dexamethasone 0.05% (Experimental): Tobramycin 0.3%/Dexamethasone 0.05% 1 drop 4 times daily in both eyes
  Interventions: Drug: Tobramycin 0.3%/Dexamethasone 0.05%
- TOBRADEX (Active Comparator): TOBRADEX 1 drop 4 times daily in both eyes
  Interventions: Drug: TOBRADEX

INTERVENTIONS:
Drug: Tobramycin 0.3%/Dexamethasone 0.05% — Tobramycin 0.3%/Dexamethasone 0.05% 1 drop in both eyes 4 times daily for at least 3 days
  Arms: Tobramycin 0.3%/Dexamethasone 0.05%
Drug: TOBRADEX — TOBRADEX 1 drop in both eyes 4 times daily for at least 3 days
  Arms: TOBRADEX

SUMMARY:
The purpose of this study is to describe the differences in efficacy between TOBRADEX Ophthalmic Suspension and Tobramycin 0.3%/Dexamethasone 0.05% Ophthalmic Suspension in the treatment of ocular inflammation and infection associated with blepharaconjunctivitis

ELIGIBILITY:
Inclusion Criteria:

* Ocular inflammation associated with blepharaconjunctivitis

Exclusion Criteria:

* ocular allergy
* ocular disorders that would preclude safe administration of test article

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2007-10; Primary Completion 2008-02 (Actual); Study Completion 2008-03

CONTACTS AND LOCATIONS:
Overall Officials: Michael Brubaker, BSN MPH, Study Director — Alcon Research
Locations (1):
- Houston, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 enrolling sites (private ophthalmology clinical offices) with first subject enrolled 10/29/07 and last subject enrolled 2/14/08)
Pre-assignment Details: Parallel, 1:1 ratio; double-masked
Groups:
- Tobramycin 0.3%/Dexamethasone 0.05%: Tobramycin 0.3%/Dexamethasone 0.05%
- TOBRADEX Ophthalmic Suspension: TOBRADEX Ophthalmic Suspension
Period: Overall Study
Arm/Group | Tobramycin 0.3%/Dexamethasone 0.05% | TOBRADEX Ophthalmic Suspension
Started | 109 | 112
Completed | 108 | 111
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tobramycin 0.3%/Dexamethasone 0.05% | TOBRADEX Ophthalmic Suspension | Total
Number analyzed (Participants) | 109 | 112 | 221
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 2 | 6
  Between 18 and 65 years | 65 | 62 | 127
  >=65 years | 40 | 48 | 88
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 65 | 118
  Male | 56 | 47 | 103

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients Who Display Microbiological Success (Eradication of Baseline Pathogens at Day 4)
Description: Microbiological success was declared if the pre-therapy pathogens were eradicated at the Exit Visit; conversely, microbiological failure was declared if pre-therapy pathogens persisted at the exit visit. The microbiological outcomes were calculated based on an algorithm that assessed whether pre-therapy pathogens were eradicated or persisted as demonstrated by comparative characterization of recovered bacteria.
Time Frame: Day 4 - Test Of Cure (TOC) compared to Day 0
Measure: Number; unit: Percent of patients
Arm/Group | Tobramycin 0.3%/Dexamethasone 0.05% | TOBRADEX Ophthalmic Suspension
Number analyzed (Participants) | 109 | 112
Percent of patients | 100.0 | 94.4

ADVERSE EVENTS:
Arm/Group | Tobramycin 0.3%/Dexamethasone 0.05% | TOBRADEX Ophthalmic Suspension
Serious Adverse Events (participants affected / at risk) | 0/109 | 0/112
Other Adverse Events (participants affected / at risk) | 0/109 | 0/112

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor is allowed 30 days to review publication. With reasonable justification, sponsor may require the publication to be withheld an additional 60 days to obtain patent protection. Sponsor may request deletion of any trade secret, proprietary, or confidential information.